CLINICAL TRIAL: NCT04637646
Title: Evaluation of Cardiac Affections in Patients With Mucopolysaccharidosis (MPS) in Assuit University Children Hospital (AUCH)
Acronym: MPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Rageh Dardiry, researcher, Assiut University
Other Study IDs: cardiac affections in MPS
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Mucopolysaccharidoses
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with MPS

SUMMARY:
This study aims to evaluate the different cardiac changes in the various types of MPS disorder and define the outcome of these cardiac abnormalities in those patients admitted to assuit University Children Hospital

DETAILED DESCRIPTION:
The mucopolysaccharidoses (MPSs) are inherited lysosomal storage disorders caused by the absence of functional enzymes that contribute to the degradation of glycosaminoglycans (GAGs). The progressive systemic deposition of GAGs results in multi-organ system dysfunction that varies with the particular GAG deposited and the specific enzyme mutation(s) present.

Cardiac involvement has been reported in all MPS syndromes and is a common and early feature, particularly for those with MPS I, II, and VI. Cardiac valve thickening, dysfunction (more severe for left-sided than for right-sided valves), and hypertrophy are commonly present; conduction abnormalities, coronary artery and other vascular involvement may also occur. Cardiac disease emerges silently and contributes significantly to early mortality. The clinical examination of individuals with MPS is often difficult due to physical and, sometimes, intellectual patient limitations. The absence of precordial murmurs does not exclude the presence of cardiac disease. Echocardiography and electrocardiography are key diagnostic techniques for evaluation of valves, ventricular dimensions and function.

ELIGIBILITY:
Inclusion Criteria:

- All the patients at any age up to 18 years with any type of MPS confirmed by the enzymatic assay

Exclusion Criteria:

* any patient other than MPS

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients with mucopolysacchridosis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-29 (Estimated); Study Completion 2022-01-29 (Estimated)

PRIMARY OUTCOMES:
Rate of Cardiac affection in patients with MPS | on enrollment
  cardiac affection in MPS patients